CLINICAL TRIAL: NCT01760161
Title: A Randomised, Double-blind Study to Evaluate the Effect of Bilateral Dual Transversus Abdominis Plane Block on Postoperative Pain and Plasma Concentration of Ropivacaine After Robotic Assisted Laparoscopic Surgery
Brief Title: Bilateral Dual Transversus Abdominis Plane Block for Robotic Assisted Laparoscopic Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No signal on pain-score
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Nils Bjerregaard, Consultant Anestetist, Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20120042
Record Dates: First submitted 2012-12-19; First posted 2013-01-04 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Pain Treatment; Robotic Assisted Laparoscopic Surgery; Bilateral Dual Transversus Abdominis Plane Block
Keywords: postoperative pain; opioid consumption; termanalgesia; plasmaropivacain level
MeSH Terms: conditions — Agnosia; Pain, Postoperative | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ropivacain (Active Comparator): Ropicacain 3,75 mg/ml 15 ml x 4 when placing the Bilateral Dual Transverus Abdominis Plane block
  Interventions: Drug: Ropivacaine
- Isotonic potassium chloride (Placebo Comparator): Isotonic potassium chloride 15 ml x 4 when placing the bilateral dual transverus abdominis plane block.
  Interventions: Drug: Isotonic potassium chloride

INTERVENTIONS:
Drug: Ropivacaine — Ropicacain 3,75 mg/ml 15 ml x 4 when placing the Bilateral Dual Transverus Abdominis Plane block
  Arms: Ropivacain
Drug: Isotonic potassium chloride — Isotonic potassium chloride 15 ml x 4 when placing the bilateral dual transverus abdominis plane block.
  Arms: Isotonic potassium chloride

SUMMARY:
To evaluate the effects of bilateral dual transversus abdominis plane block on postoperative pain after robotic assited laparoskopic surgery and measure the plasma-level of ropivacain after the bilateral dual transversus abdominis plane block.

DETAILED DESCRIPTION:
After randomisation patients for robotic assisted laparoscopic surgery will receive bilateral dual transversus abdominis plane block containing either ropivacain or isotonic potassium chloride.

The investigators will record pain-score, opioid-consumption and sensibility on the abdominal wall in the postoperative periode.

Also a blood sample will be taken at 15, 30, 60, 120 and 240 minutes after the block in order to measure the plasma-level of ropivacain after bilateral dual transversus abdominis plane block.

The investigators assume that there will be significant effect on postoperative pain and that the level of plasma-ropivacain will be acceptable.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for robotic assisted laparoscopis surgery
* acceptance to participate

Exclusion Criteria:

* allergies to local analgetics
* daily use of strong opioids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-12 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Pain-score on numerical rating scale | 4 hours after surgery

SECONDARY OUTCOMES:
Administration of opioids | The first 24 hours after surgery.
Pain-score on numerical rating scale | 8 hours after surgery
Pain-score on numerical rating scale | 24 hours after surgery

OTHER OUTCOMES:
Thermoanalgesia at dermatome-level th6-th12 | 1 hour after bilateral dual transversus abdominis plane block
Plasma-ropivacain level | 15, 30, 60, 120 and 240 mins after the block

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg Hospital, Aalborg, Region Nord, Denmark